CLINICAL TRIAL: NCT07021131
Title: Continuous Serratus Posterior Plane Block Versus Continuous Erector Spine Plane Block for Video-assisted Thoracoscopic Surgery: a Prospective Randomized Non-inferiority Trial
Brief Title: Serratus Posterior Plane Block vs Erector Spine Plane Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s. (Other)
Responsible Party: Principal Investigator, Daniel Nalos, senior researcher, Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SERRATUS
Record Dates: First submitted 2025-05-19; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Regional Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block (No Intervention): Patients undergoing VATS with the use of continuous peripheral nerve block type A.
- Serratus Posterior Plane Block (Experimental): Patients undergoing general anaesthesia with continuous peripheral block type B.
  Interventions: Procedure: new type of peripheral block Serratus Posterior Plane Block

INTERVENTIONS:
Procedure: new type of peripheral block Serratus Posterior Plane Block — Intervention will be Serratus Posterior Plane Block.
  Arms: Serratus Posterior Plane Block

SUMMARY:
Analgesia related to the administration of local anesthetic solution into the fascia of erector spinae muscle is mediated by the effect of local anesthetic on the posterior and lateral branches of the anterior part of the spinal nerve. Comparable analgesic efficiency after the administration of both nerve blocks would reject the widespread theory of the paravertebral site of effect of the local anesthetic in ESPB.

ELIGIBILITY:
Inclusion Criteria:

* Patiens undergoing VATS-surgery

Exclusion Criteria:

* Age < 20 years
* Body Mass Index >35 kg/m2
* Technical difficulties with the nerve block administration and/or subsequent bolus application
* Abnormal course of the surgery (e.g. conversion to thoracotomy) or the postoperative phase (e.g. surgical revision of the chest)
* Patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid dose in 72 hours | from end of surgery to 72 hours after the end surgery
  Irrespective of the type of the block, 20 mls of 0.25 % bupivacaine will be administered to the block catether every 8 hours. Every patients will receive non-opioid analgesics according to standardized ward guideline. VAS score is recorded at least every 3 hours (except for time patient is asleep). Any time patient reports VAS score >=5, he/she will receive 5 mg of morphine intravenously (or equivalent dose of Oxycodone per os). Cumulative dose of opioids will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslava Korfova, Principal Investigator — Krajská zdravotní, a.s. - Masarykova nemocnice v Ústí nad Labem, o.z.
Locations (1):
- Krajská zdravotní, a.s. - Masarykova nemocnice v Ústí nad Labem, o.z., Ústí nad Labem, Ústecký kraj, Czechia

IPD SHARING:
Plan to Share IPD: Undecided